CLINICAL TRIAL: NCT05132205
Title: Radiofrequency Ablation of Papillary Thyroid Microcarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: RF Medical Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00236242
Record Dates: First submitted 2021-11-10; First posted 2021-11-24 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Papillary Thyroid Cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiofrequency Ablation (Experimental): Patients will receive RFA as a one-time intervention, with a possible second treatment after 6 months if adequate resolution is not noted on ultrasound.
  Interventions: Procedure: Radiofrequency Ablation

INTERVENTIONS:
Procedure: Radiofrequency Ablation — Radiofrequency Ablation using RFMedical device.

SUMMARY:
Traditionally, surgery has been the standard recommendation for treating papillary thyroid cancer. The risk of surgery including permanent hoarseness, permanent hypocalcemia, a mid-cervical scar, and the potential for permanent hypothyroidism may be unacceptable for some patients, especially with low risk papillary thyroid carcinoma. The recent American Thyroid Association guidelines have proposed the option of active surveillance with low risk papillary thyroid cancer less than 210 mm. However, most patients find observation anxiety provoking knowing of having cancer. Radiofrequency ablation (RFA) of small low risk papillary thyroid cancer is a promising therapeutic modality for these patients that reduces the risks associated with surgery and the anxiety of taking a watchful approach. However, this technique has not been validated in the North American population.

The investigators aim to describe the investigators' initial experience with RFA of low risk papillary thyroid microcarcinoma (PTMC) compared to active surveillance (AS) done by Head and Neck Endocrine surgeons at Johns Hopkins Medical Institute.

Primary objective:

* To evaluate the safety, efficacy and oncological outcomes of the procedure.

Secondary objective:

* To determine the patient functional outcomes in comparison to the observational control.

ELIGIBILITY:
Inclusion Criteria:

* All patients regardless of sex or race between the ages 18-100 with biopsy proven PTMC with a Bethesda V or VI pathology or indeterminate cytology on fine-needle aspiration cytology (FNAC) who are recommended for treatment (Bethesda III/IV).
* Solitary thyroid nodule <20mm in maximal dimension.
* No sonographic evidence of extrathyroidal invasion, lymph node metastases, or distant metastases.
* There must be at least 1 mm of normal tissue as a margin, without sonographic evidence of contact with the capsule.

Exclusion Criteria:

* Patients with other histological types of thyroid malignancy other than papillary thyroid cancer such as medullary carcinoma, Proto-oncogene serine/threonine kinase (BRAF) or Telomerase reverse transcriptase (TERT) mutations
* Clinically apparent multicentricity
* Lesions larger than 20 mm in maximum diameter.
* Recurrent laryngeal nerve palsy.
* Extension of nodule to posterior thyroid capsule.
* Ultrasound or other imaging studies revealing cervical lymph node involvement or distant metastases.
* Pregnancy.
* Pacemaker.
* Previous RFA.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Percentage change in nodule volume | Baseline and 12 months
  This will assess the percentage change in nodule volume (cubic millimeters).

SECONDARY OUTCOMES:
Percentage change in nodule volume | Baseline and 6 months
  This will assess the percentage change in nodule volume (cubic millimeters).
Percentage change in nodule volume | Baseline and 24 months
  This will assess the percentage change in nodule volume (cubic millimeters).
Change in voice related quality of life as assessed by the VHI-10 | Baseline and 6 months
  Change from baseline in Voice Handicap index (VHI-10) score. Score ranges from 0-40. Higher score indicates worse symptoms.
Change in voice related quality of life as assessed by the VHI-10 | Baseline and 12 months
  Change from baseline in the VHI-10 score. Score ranges from 0-40. Higher score indicates worse symptoms.
Change in voice related quality of life as assessed by the VHI-10 | Baseline and 24 months
  Change from baseline in the VHI-10 score. Score ranges from 0-40. Higher score indicates worse symptoms.
Scar cosmesis score | 6 months
  Average score on Scar cosmesis assessment and rating (SCAR) scale. Score ranges from 0-15. Higher score indicates worse scar.
Scar cosmesis score | 12 months
  Average score on SCAR scale. Score ranges from 0-15. Higher score indicates worse scar.
Scar cosmesis score | 24 months
  Average score on SCAR scale. Score ranges from 0-15. Higher score indicates worse scar.
Change in eating assessment score as assessed by the EAT-10 | Baseline and 6 months
  Change from baseline on Eating assessment tool (EAT-10) score. Score ranges from 0-40. Higher score indicates worse symptoms.
Change in eating assessment score as assessed by the EAT-10 | Baseline and 12 months
  Change from baseline on EAT-10 score. Score ranges from 0-40. Higher score indicates worse symptoms.
Change in eating assessment score as assessed by the EAT-10 | Baseline and 24 months
  Change from baseline on EAT-10 score. Score ranges from 0-40. Higher score indicates worse symptoms.
Change in overall quality of life assessed by the PROMIS score | Baseline and 6 months
  Change from baseline on Patient-Reported Outcomes Measurement Information System (PROMIS)-29 score. Score ranges from 0-100. Higher score indicates worse symptoms.
Change in overall quality of life assessed by the PROMIS score | Baseline and 12 months
  Change from baseline on PROMIS-29 score. Score ranges from 0-100. Higher score indicates worse symptoms.
Change in overall quality of life assessed by the PROMIS score | Baseline and 24 months
  Change from baseline on PROMIS-29 score. Score ranges from 0-100. Higher score indicates worse symptoms.
Number of complications | 12 months
  Counts of skin burn, hematoma and vocal cord palsy.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Russell, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No